CLINICAL TRIAL: NCT01705015
Title: Organ Transplantation Rehabilitation: Effect of Bedside Exercise Device and Activity Reinforcement for Heart or Liver Transplantation Recipients in Early Postoperative Period
Brief Title: Organ Transplantation Rehabilitation: Effect of Bedside Exercise Device and Activity Reinforcement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NSC101-2314-B-002-006-MY3
Record Dates: First submitted 2012-09-11; First posted 2012-10-12 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-09

CONDITIONS: Heart Transplantation; Liver Transplantation
Keywords: exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- UCFit plus direct feedback about exercise (Experimental): Subjects assigned to higher feedback will be encouraged to look at the summary of daily data about pedaling and will be encouraged to progress activity - more repetitions per minute (RPM range from 10-60), more frequent sessions (up to 3 times daily), longer sessions (from 5-20 minutes), and exertion against larger forces (no resistance, mild, moderate) for the legs. These subjects will also be encouraged to carry out pedaling with the upper extremities once a day, if the arms are free of lines that could be damaged. Progression of leg exercises would be within the capability and motivation of each subject, but would not exceed increments of 10% from one day to the next in any one of these parameters. Graphical displays that can be used for feedback will be available at the patient's bedside. The staff, patient and family will be able to view these bar graphs.
  Interventions: Behavioral: direct feedback about exercise
- UCFit plus encouraged exercise (Placebo Comparator): These subjects will receive a graph of the total number of minutes cycled each day and the average RPMs. The coordinator will only encourage these subjects to try to increase their total cycling time. These bar graphs will not be posted, but will be left by the bedside.
  Interventions: Behavioral: PLacebo

INTERVENTIONS:
Behavioral: direct feedback about exercise
  Arms: UCFit plus direct feedback about exercise
Behavioral: PLacebo — UCFit plus encouraged exercise
  Arms: UCFit plus encouraged exercise

SUMMARY:
The aims of this 3-year randomized, single-blinded clinical trial are to compare the effect of high and low feedback about performance on the bedside exercise device in heart or liver transplantation recipients during the hospitalization immediately after transplantation. The hypotheses of the study are heart/liver transplantation recipients who have high feedback about performance on the bedside exercise device will progressively increase their level of exercise over the course of their hospitalization, more independent in ambulation level, better walking speed and 6-minute walk test at discharge, and better cardiorespiratory fitness at 4-8 weeks after transplantation than those who receive low feedback. The adult patients who newly receive heart or liver transplantation at National Taiwan University Hospital will be evaluated for eligibility of the study in the acute postoperative period. The study will be conducted in both the intensive care unit and ward environments. The study subjects will be randomized to either high or low feedback about performance on the bedside exercise device which uses hand/foot pedals that record exerted forces against adjustable resistances, measure repetitions of upper and lower extremity cycling movements, and give feedback about performance via a wireless internet connection. The study will also monitor the amount of daily movement activity of all subjects in this trial by using triaxial accelerometers, and the activity recognition algorithms developed by engineers and computer scientists at University of California Los Angeles. The outcome measures include level of independence for walking, walking speed, 6-minute walk test, and cardiopulmonary exercise testing by the blinded observers. The study expects to enroll at least 50 heart transplantation recipients and 60 liver transplantation recipients in 3 years. The results of this study will offer much insight into activity levels of heart or liver transplantation recipients during early postoperative period. Besides, heart transplantation recipients will receive routine phase I cardiac rehabilitation program by the physical therapists during the study but not liver transplantation recipients. We might be able to evaluate the interaction effects of routine physical therapy and UCFit exercise among our study subjects. Our data will also provide insight into just how active or inactive transplantation recipients may be and help generate ideas of organ transplantation rehabilitation program to increase their fitness-related activity prior to discharge.

ELIGIBILITY:
Inclusion Criteria:

* just received heart or liver transplantation at National Taiwan University Hospital during admission
* over age 18 years old
* living and walking independently, based on the Functional Independence Measure of activities of daily living, within 6 weeks prior to admission
* no major contraindication to participating in light-to-moderate exertion and Per their primary physician in the hospital
* be able to follow and retain 3 minutes later verbal directions to carry out a simple upper and a lower extremity repetitive exercise, such as leg lifts.

Exclusion Criteria:

* unlikely to survive for 3 months
* body mass index >30
* progressive decline in medical status by symptoms or laboratory data (e.g., new onset renal failure or transplant rejection) at the time of entry that is likely to interfere with exercise capacity (subjects may participate once stable);
* skin breakdown that will interfere with positioning for exercise
* inability to lift each leg so that the heel is 6 inches above the bed
* cardiopulmonary contraindication to modest exercise per the care team, such as angina, deep vein thrombosis or hypoxia
* fractures or contractures that prevent use of an extremity for pedaling
* A hemiparesis that is mild enough to permit voluntary placement of the hand and foot onto the apparatus will not be an exclusion, but lesser motor control will.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
A.Level of independence for walking 150 feet and the ratio of subjects who achieve independence in walking 150 feet. B. Walking speed for 50 feet. C. 6-minute walk test. D. Findings of cardiopulmonary exercise testing | At discharge of hospital stay, an expected average of 5 weeks, up to 8 weeks after transplantation
  A.* Level of independence for walking 150 feet (or only for 50 feet if that is feasible) and the ratio of subjects who achieve independence in walking 150 feet in each group based on the criteria of the 7-level scale; B.* Walking speed for 50 feet (or for a subject's lesser feasible distance);C.* 6-minute walk test (including the walking distance in 3 and 6 minutes); D.* Peak oxygen uptake of cardiopulmonary exercise testing (if the exercise testing is not feasible at discharge, findings within 8 weeks after transplantation will be acceptable)

SECONDARY OUTCOMES:
A.Total amount of exercise. B.Short Form-36. C. Length of stay in the intensive care unit and hospital. D.Rate of rehospitalization. E.Adverse responses and complications related to exercise. | At discharge of hospital stay, an expected average of 5 weeks, up to 8 weeks after transplantation, and 30 days after discharge
  A.* Total number of daily sessions and total minutes of exercise during the hospital stay; B.* Health-related quality of life by Short Form-36 questionnaire; C.* Length of stay in the intensive care unit and hospital post transplantation; D.* Rate of rehospitalization within 30 days of discharge; E.* Adverse responses and complications related to exercise.

CONTACTS AND LOCATIONS:
Overall Officials: SSU-YUAN CHEN, MD PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan